CLINICAL TRIAL: NCT04625309
Title: Adaptive Sports for Individuals With a Physical Disability: Impact on the ICF Domains
Brief Title: Effect of Adaptive Sports After Acquired Physical Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPORT DISABILITY
Record Dates: First submitted 2020-02-20; First posted 2020-11-12 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Spinal Cord Injuries; Sports Physical Therapy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sport (Experimental): This group will be made up of subjects with a spinal cord injury that are actively participating in adaptive sports teams.
  Interventions: Other: Adaptive sports
- No sport (No Intervention): This group will be made up of subjects with a spinal cord injury that are not actively participating in any sports team.

INTERVENTIONS:
Other: Adaptive sports — This will be the number of hours per week the subjects actively partake in adaptive sports teams.
  Arms: Sport

SUMMARY:
This study is a cross-sectional trial which aims to evaluate the effect of practicing a physical activity on different domains of the ICF among individuals with an acquired physical disability. Two different groups of individuals with a spinal cord injury will be enrolled: one composed of subjects who manage to reach the WHO's recommendations regarding physical activity, and the other of subjects who do not.

DETAILED DESCRIPTION:
The present study will recruit participants based on a set of defined eligibility criteria, in adaptive sports clubs teams and in groups or associations of individuals with an acquired, and permanent, physical disability. Based on the presence or absence of a regular physical activity practice undertaken by the subjects who give their consent to participate in the study, they will be divided into two groups: one where individuals regularly practice a physical activity, and one where they do not.

A set of defined outcome measures (detailed in the "Outcome Measures"section) will be assessed in both groups.

The outcomes measures will be analysed statistically, using SPSS software. Depending on the nature of the variables (qualitative or quantitative), different tests will be performed. Normality will also be verified and will determine which statistical analysis will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed non-progressive spinal cord injury
* dependent on wheelchair for mobility
* more than 6 months since diagnosis of spinal injury
* able to understand and speak french

Exclusion Criteria:

* medical contra-indication to the testing
* cognitive deficiency which limits communication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Pain experienced during mobility | Throughout the study, an average of 4 months
  This variable will be measured through a Likert scale out of 5, where greater values show more pain during mobility. Subjects will be asked to rate presence, frequency and intensity of pain felt in the upper-limb when wheeling in their daily environments.
Fatigue Severity | Throughout the study, an average of 4 months
  This variable will be measured using a validated questionnaire, "Fatigue Severity scale". The minimum score is 9, and the maximum is 63. The higher the score, the greater the fatigue severity (= worse outcome for the participant).
Independence in mobility of daily living | Throughout the study, an average of 4 months
  This variable will be measured using the validated "Spinal Cord Independence Measure -mobility". Minimum score is 0 while maximum score is 40. The higher the score, the better the independence of the participant (=better outcome).
Physical activity level | Through study completion, an average of 4 months
  Measured by a validated questionnaire, "Physical Activity Scale for Individuals with a Physical Disability".
Social participation | Throughout the study, an average of 4 months
  This variable will be measured through the validated "Reintegration to Normal Living" index. Minimum score is 0, maximum score is 100. The higher the score, the better the outcome.
Quality of Life: WHOQOL-BREF | Throughout the study, an average of 4 months
  This variable will be measured through the World Health Organization's 8th version questionnaire, the WHOQOL-BREF. Every one of the 4 domain can obtain a score ranging from 0 (minimum) to 100 (maximum). The higher the score, the greater the quality of life.
patient's medical history | Throughout the study, an average of 4 months
  We will ask the subjects to report how many times they were hospitalised in the last six months and how many times they experienced a serious health-complication. We will also ask them how many times per week they receive physiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Declerck, PT, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Université catholique de Louvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No